CLINICAL TRIAL: NCT06627257
Title: A Phase 1b, Double-Blind, Randomized, Placebo-Controlled, Antigen Dose-Escalation Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of LEP-F1 + GLA-SE in Healthy Adult Participants in Areas Endemic for Leprosy
Brief Title: Trial LEP-F1 + GLA-SE in Healthy Adult in Areas Endemic for Leprosy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Oswaldo Cruz Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ASCLIN 001/2023
Record Dates: First submitted 2023-08-21; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-01

CONDITIONS: Leprosy
MeSH Terms: conditions — Leprosy | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Participants, investigators, study personnel performing any study-related assessments following study injection, and laboratory personnel performing immunology assays will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LepVax (Experimental): Participants will be randomized within each Group to receive three doses of vaccine administered IM on Days 0, 28, and 56. Participants will be monitored for one year following the last study injection, including safety laboratory analyses 7 days following each study injection. Blood samples will be obtained for immunological assays at Days 0, 35, 63, and 168.
  Interventions: Drug: LepVax (2 μg LEP-F1 + 5 μg GLA-S): Low dose; Drug: LepVax (10 μg LEP-F1 + 5 μg GLA-SE): High dose
- Placebo groups (Placebo Comparator): Participants will be randomized within each Group to receive three doses of placebo administered IM on Days 0, 28, and 56. Participants will be monitored for one year following the last study injection, including safety laboratory analyses 7 days following each study injection. Blood samples will be obtained for immunological assays at Days 0, 35, 63, and 168.
  Interventions: Other: Placebo Comparator: Placebo

INTERVENTIONS:
Drug: LepVax (2 μg LEP-F1 + 5 μg GLA-S): Low dose — 2 μg LEP-F1 + 5 μg GLA-SE will be administered by IM injection on Days 0,28, and 56 in healthy participants.
  Other Names: LepVax
  Arms: LepVax
Drug: LepVax (10 μg LEP-F1 + 5 μg GLA-SE): High dose — 10 μg LEP-F1 + 5 μg GLA-SE will be administered by IM injection on Days 0,28, and 56 in healthy participants.
  Other Names: LepVax
  Arms: LepVax
Other: Placebo Comparator: Placebo — Sterile normal saline for injection will be administered by IM injection on Days 0, 28, and 56 in healthy participants and paucibacillary leprosy patients.
  Other Names: Sterile normal saline for injection.
  Arms: Placebo groups

SUMMARY:
This is a phase 1b, double-blind, randomized, placebo-controlled clinical trial to evaluate the safety, tolerability, and immunogenicity of LEP-F1 + GLA-SE compared to placebo administered as three intramuscular (IM) injections in adult participants aged 18 to 55.

DETAILED DESCRIPTION:
The LepVax Clinical Development Plan includes two indications for use. The first would be the prophylactic indication, where individuals at greater risk, such as contacts of patients affected by leprosy and who may be subclinically infected with M. leprae, would be vaccinated. This concept is not unique and many countries, such as Brazil, re-immunize leprosy patients and their close contacts with BCG (5, 12, 13). The proposed clinical trial, however, is to establish an initial safety profile in a leprosy endemic region where healthy adults will be included. The second use indication is for therapeutic indication of the vaccine that would be an adjuvant to the current treatment for leprosy. After vaccine safety is established, phase 2 protocols in leprosy patients will be proposed to assess vaccine dose and safety in this population, and then move on to phase 3, where vaccine efficacy will be evaluated.

This phase 1b, double-blind, randomized, placebo-controlled clinical trial will evaluate the safety, tolerability, and immunogenicity of LEP-F1 + GLA-SE in healthy adults. Two dose levels of LEP-F1 will be tested (2 and 10 µg of LEP-F1) and a fixed dose of 5 µg of GLA-SE in adults. These doses were selected because they demonstrated an acceptable safety and immunogenicity profile in the LEPVPX-118 study, the first clinical trial in humans. This study will establish a safety and immunogenicity profile in an endemic population that will allow the vaccine to advance in clinical development.

Participants will be randomized within each Group to receive three doses of vaccine or placebo administered IM on Days 0, 28, and 56. Participants will be monitored for one year following the last study injection, including safety laboratory analyses 7 days following each study injection. Blood samples will be obtained for immunological assays at Days 0, 35, 63, and 168.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 55 years old.
* They should be in good general health, confirmed by a medical history and physical examination, with negative clinical evaluation for leprosy.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on study vaccination days (D0, D28, and D56). They must not be breastfeeding and must use at least one method of contraception from the time of study enrollment (Day 0) through 30 days after the last injection if they have sex with men.
* Screening laboratory tests with normal, within laboratory reference limits for: sodium, potassium, AST, ALT, total bilirubin, alkaline phosphatase, creatinine, glucose, total WBC count, hemoglobin and platelet count. Abnormal results may be repeated at the discretion of the Principal Investigator and/or sub-investigators, who may share doubts with the sponsor's Scientific Leader and if necessary, with the DSMB.
* Negative serological tests for: HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
* Normal or not clinically significant urinalysis as determined by the study doctor or designee. Abnormal results may be repeated at the discretion of the Principal Investigator.
* Must be able to complete the study adverse events diary.
* Must consent to participate in the study, be able and willing to make all evaluation visits, be accessible by telephone or home visits, and live in the region until study follow-up completion.
* Having completed the primary vaccination course for Covid 19, at least 14 days before inclusion in the study. If 14 days have not been completed, the participant may be rescheduled for a new eligibility assessment

Exclusion Criteria:

* History of infection with Mycobacterium leprae.
* History of exposure to experimental products containing GLA-SE.
* History of active tuberculosis or documented recurrence.
* History of previous infection with other non-tuberculous mycobacteria.
* Participation in another trial protocol and/or receipt of any trial products in the last 3 months prior to screening.
* Treatment with immunosuppressive drugs (eg, oral or injectable steroids such as prednisone; high-dose inhaled steroids) or cytotoxic therapies (eg, chemotherapy or radiotherapy) within six months prior to screening.
* Have received blood transfusion within the last 3 months prior to screening.
* Donated blood products (platelets, whole blood, plasma, etc.) within the last month prior to screening.
* Received any vaccine 1 month prior to screening or planned immunizations during the follow-up from D0 to D63 and D154 to D168.
* History of autoimmune disease or other immunosuppressive causes.
* History of any other uncompensated acute or chronic disease (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, hematological, metabolic or renal disease, uncontrolled hypertension) or use of medications that, in the opinion of the Principal Investigator, may interfere with safety or immunogenicity of the vaccine.
* Rash, tattoos, or any other dermatological condition that may adversely affect the injection site of the vaccine or interfere with its evaluation.
* Body mass index (BMI) ≥ 32.
* Systemic arterial hypertension (systolic > 150 or diastolic > 95).
* History of psychiatric illness with current medication use.
* Alcohol or drug abuse in the last 6 months prior to screening.
* Chronic smoker (1 pack or more per day).
* History of previous anaphylaxis or severe allergic reaction to unknown vaccines or allergens.
* Individuals who do not wish to cooperate with all procedures recommended in the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Phase 1b_The number of participants who receive the injection and experience local and systemic reactions within 7 days of each study injection. | 7 days following each injection
  The number of participants who receive the injection and experience local and systemic reactions within 7 days of each study injection.
Phase 1b_Number of participants experiencing unsolicited AEs | Day 0 to Day 84 following each injection
  The number of participants spontaneously reporting adverse events from Day 0 to Day 84.
Phase 1b_The number of physician-attended adverse events | Through study completion, an average of 1 year
  The number of physician-attended adverse events considered to be related to any of the study injections reported at any time during the study period.

SECONDARY OUTCOMES:
Phase 1b_IgG antibody responses to LEP-F1 by ELISA on Days 0, 35, 63,and 168. | Days 0, 35, 63 and 168
  IgG antibody responses to LEP-F1 by ELISA on Days 0, 35, 63, and 168
Phase 1b_ The T cell responses measured by LEP-F1-specific cytokine production in PBMC assay by ELISA or multiplex assay on Days 0, 35, 63,and 168.whole blood assay | Days 0, 35, 63 and 168
  The T cell responses measured by LEP-F1-specific cytokine production in PBMC assay by ELISA or multiplex assay on Days 0,35, 63, and 168.

OTHER OUTCOMES:
The T cell responses measured by multiparametric flow cytometry in PBMCs | Days 0,35,63 and 168
  The T cell responses measured by multiparametric flow cytometry in PBMCs on Days 0, 35, 63, and 168.
Phase 1b_The assays of candidate biomarkers measured on Day 0 and 63 including gene expression signatures and serum protein multiplex assay. | Day 0 and 63]
  The assays of candidate biomarkers measured on Day 0 and 63 including gene expression signatures and serum protein multiplex assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Oswaldo Cruz Institue, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duthie MS, Frevol A, Day T, Coler RN, Vergara J, Rolf T, Sagawa ZK, Marie Beckmann A, Casper C, Reed SG. A phase 1 antigen dose escalation trial to evaluate safety, tolerability and immunogenicity of the leprosy vaccine candidate LepVax (LEP-F1 + GLA-SE) in healthy adults. Vaccine. 2020 Feb 11;38(7):1700-1707. doi: 10.1016/j.vaccine.2019.12.050. Epub 2019 Dec 30. PMID 31899025
- [Background] Cunha SS, Alexander N, Barreto ML, Pereira ES, Dourado I, Maroja Mde F, Ichihara Y, Brito S, Pereira S, Rodrigues LC. BCG revaccination does not protect against leprosy in the Brazilian Amazon: a cluster randomised trial. PLoS Negl Trop Dis. 2008 Feb 13;2(2):e167. doi: 10.1371/journal.pntd.0000167. PMID 18270542
- [Background] Duppre NC, Camacho LA, da Cunha SS, Struchiner CJ, Sales AM, Nery JA, Sarno EN. Effectiveness of BCG vaccination among leprosy contacts: a cohort study. Trans R Soc Trop Med Hyg. 2008 Jul;102(7):631-8. doi: 10.1016/j.trstmh.2008.04.015. Epub 2008 Jun 2. PMID 18514242
- [Background] Bertholet S, Goto Y, Carter L, Bhatia A, Howard RF, Carter D, Coler RN, Vedvick TS, Reed SG. Optimized subunit vaccine protects against experimental leishmaniasis. Vaccine. 2009 Nov 23;27(50):7036-45. doi: 10.1016/j.vaccine.2009.09.066. Epub 2009 Sep 26. PMID 19786136
- [Background] Baldwin SL, Bertholet S, Kahn M, Zharkikh I, Ireton GC, Vedvick TS, Reed SG, Coler RN. Intradermal immunization improves protective efficacy of a novel TB vaccine candidate. Vaccine. 2009 May 18;27(23):3063-71. doi: 10.1016/j.vaccine.2009.03.018. Epub 2009 Mar 26. PMID 19428920
- [Background] Olugbile S, Kulangara C, Bang G, Bertholet S, Suzarte E, Villard V, Frank G, Audran R, Razaname A, Nebie I, Awobusuyi O, Spertini F, Kajava AV, Felger I, Druilhe P, Corradin G. Vaccine potentials of an intrinsically unstructured fragment derived from the blood stage-associated Plasmodium falciparum protein PFF0165c. Infect Immun. 2009 Dec;77(12):5701-9. doi: 10.1128/IAI.00652-09. Epub 2009 Sep 28. PMID 19786562
- [Background] Baldwin SL, Shaverdian N, Goto Y, Duthie MS, Raman VS, Evers T, Mompoint F, Vedvick TS, Bertholet S, Coler RN, Reed SG. Enhanced humoral and Type 1 cellular immune responses with Fluzone adjuvanted with a synthetic TLR4 agonist formulated in an emulsion. Vaccine. 2009 Oct 9;27(43):5956-63. doi: 10.1016/j.vaccine.2009.07.081. Epub 2009 Aug 11. PMID 19679214
- [Background] Global leprosy update, 2014: need for early case detection. Wkly Epidemiol Rec. 2015 Sep 4;90(36):461-74. No abstract available. English, French. PMID 26343055
- [Background] Scollard DM. The biology of nerve injury in leprosy. Lepr Rev. 2008 Sep;79(3):242-53. PMID 19009974
- [Background] Coler RN, Bertholet S, Moutaftsi M, Guderian JA, Windish HP, Baldwin SL, Laughlin EM, Duthie MS, Fox CB, Carter D, Friede M, Vedvick TS, Reed SG. Development and characterization of synthetic glucopyranosyl lipid adjuvant system as a vaccine adjuvant. PLoS One. 2011 Jan 26;6(1):e16333. doi: 10.1371/journal.pone.0016333. PMID 21298114
- [Background] Merle CS, Cunha SS, Rodrigues LC. BCG vaccination and leprosy protection: review of current evidence and status of BCG in leprosy control. Expert Rev Vaccines. 2010 Feb;9(2):209-22. doi: 10.1586/erv.09.161. PMID 20109030
- [Background] Setia MS, Steinmaus C, Ho CS, Rutherford GW. The role of BCG in prevention of leprosy: a meta-analysis. Lancet Infect Dis. 2006 Mar;6(3):162-70. doi: 10.1016/S1473-3099(06)70412-1. PMID 16500597
- [Background] Wilder-Smith EP, Van Brakel WH. Nerve damage in leprosy and its management. Nat Clin Pract Neurol. 2008 Dec;4(12):656-63. doi: 10.1038/ncpneuro0941. Epub 2008 Nov 11. PMID 19002133
- See also: Scollard DM. The biology of nerve injury in leprosy. Lepr Rev 2008; 79:242-53. — https://pubmed.ncbi.nlm.nih.gov/19009974/
- See also: Wilder-Smith EP, Van Brakel WH. Nerve damage in leprosy and its management. Nature clinical practice. Neurology 2008; 4:656-63. — https://www.researchgate.net/publication/23466585_Nerve_damage_in_leprosy_and_its_management
- See also: OMS. 2015. Global leprosy update, 2014: need for early case detection. Wkly Epidemiol Rec 2014; 90:461-74. — https://www.who.int/publications/i/item/who-wer9036
- See also: Setia MS, Steinmaus C, Ho CS, Rutherford GW. The role of BCG in prevention of leprosy: a meta-analysis. Lancet Infect Dis 2006; 6:162-70. — https://www.scielo.br/j/rimtsp/a/9RLy8qtHTSfdYWSfKXKr8rc/
- See also: Merle CS, Cunha SS, Rodrigues LC. BCG vaccination and leprosy protection: review of current evidence and status of BCG in leprosy control. Expert review of vaccines 2010;9: 209-22 — https://www.ncbi.nlm.nih.gov/books/NBK78956/
- See also: Coler RN, Bertholet S, Moutaftsi M, et al. Development and characterization of synthetic glucopyranosyl lipid adjuvant system as a vaccine adjuvant. PLoS One 2011; 6: e16333 — https://pubmed.ncbi.nlm.nih.gov/21298114/
- See also: Olugbile S, Kulangara C, Bang G, et al. Vaccine potentials of an intrinsically unstructured fragment derived from the blood stage-associated Plasmodium falciparum protein PFF0165c. Infect Immun 2009; 77:5701-5709 — https://pubmed.ncbi.nlm.nih.gov/19786562/
- See also: Baldwin SL, Bertholet S, Kahn M, et al. Intradermal immunization improves protective efficacy of a novel TB vaccine candidate. Vaccine 2009; 27:3063-3071 — https://pubmed.ncbi.nlm.nih.gov/19428920/
- See also: Bertholet S, Goto Y, Carter L, et al. Optimized subunit vaccine protects against experimental leishmaniasis. Vaccine 2009; 27:7036-7045 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2783536/
- See also: Duppre NC, Camacho LA, da Cunha SS, et al. Effectiveness of BCG vaccination among leprosy contacts: a cohort study. Trans R Soc Trop Med Hyg 2008; 102:631- 8 — https://pubmed.ncbi.nlm.nih.gov/18514242/
- See also: Cunha SS, Alexander N, Barreto ML, et al. BCG Revaccination Does Not Protect Against Leprosy in the Brazilian Amazon: A Cluster Randomised Trial. PLoS Negl Trop Dis 2008; 2: e167 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2238709/
- See also: Duthie MS, Frevol A, Day T, Coler RN, Vergara J, Rolf T, et al. A phase 1 antigen dose escalation trial to evaluate safety, tolerability and immunogenicity of the leprosy vaccine candidate LepVax (LEP-F1 + GLA-SE) in healthy adults. Vaccine. 11 de fev — https://pubmed.ncbi.nlm.nih.gov/31899025/